CLINICAL TRIAL: NCT05741450
Title: A Clinical Comparison of Two Soft Contact Lenses (Iteration Under Umbrella Protocol C19-678)
Brief Title: A Clinical Comparison of Two Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: C22-724 (EX-MKTG-138)
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-02

CONDITIONS: Myopia; Hyperopia
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Intervention Model Description: All participants received Lens 1 and then Lens 2 in fixed-sequence order.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens 1 (Experimental): All participants wore Lens 1 for 15 minutes (Period 1)
  Interventions: Device: Lens 1 (monthly replacement)
- Lens 2 (Experimental): All participants wore Lens 2 for 15 minutes (Period 2)
  Interventions: Device: Lens 2 (daily disposable)

INTERVENTIONS:
Device: Lens 1 (monthly replacement) — Monthly replacement spherical silicone hydrogel contact lens for 15 minutes
  Arms: Lens 1
Device: Lens 2 (daily disposable) — Daily disposable spherical silicone hydrogel contact lens for 15 minutes
  Arms: Lens 2

SUMMARY:
The study objective was to gather short-term clinical performance data for two soft contact lenses.

DETAILED DESCRIPTION:
The aim of this subject-masked, non-randomized, controlled non-dispensing study was to evaluate the short-term clinical performance of a monthly sphere contact lens when compared to a daily disposable contact lens after 15 minutes of daily wear each.

ELIGIBILITY:
Inclusion Criteria:

* They are of legal age (18) and capacity to volunteer.
* They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
* They are willing and able to follow the protocol.
* They currently wear soft contact lenses, or have done so within the past two years.
* They are expected to be able to be fitted with the study lenses within the power range available.

Exclusion Criteria:

* They have an ocular disorder which would normally contra-indicate contact lens wear.
* They have a systemic disorder which would normally contra-indicate contact lens wear.
* They are using any topical medication such as eye drops or ointment.
* They are aphakic.
* They have had corneal refractive surgery.
* They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
* They are pregnant or lactating.
* They have an eye or health condition including an immunosuppressive or infectious disease which would, in the opinion of the investigator, contraindicate contact lens wear or pose a risk to study personnel; or a history of anaphylaxis or severe allergic reaction.
* They have taken part in any contact lens or care system clinical research within two weeks prior to starting this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Morgan, PhD, MCOptom, Principal Investigator — Eurolens Research
Locations (1):
- Eurolens Research, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Lens 1 (Monthly Replacement): All participants wore Lens 1 for 15 minutes (Period 1)
- Lens 2 (Daily Disposable): All participants wore Lens 2 for 15 minutes (Period 2)
Period: Period 1: Lens 1, 15 Minutes
Arm/Group | Lens 1 (Monthly Replacement) | Lens 2 (Daily Disposable)
Started | 45 | 0 (All participants received Lens 1 in Period 1.)
Completed | 45 | 0
Not Completed | 0 | 0
Period: Period 2: Lens 2, 15 Minutes
Arm/Group | Lens 1 (Monthly Replacement) | Lens 2 (Daily Disposable)
Started | 0 (All participants received Lens 2 in Period 2.) | 45
Completed | 0 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: All participants who participated in the clinical trial.
Arm/Group | Overall Study
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age data is presented as stratified by the sex of the participant
  years
    Female: number analyzed (Participants) | 28
    Female | 32.4 (11.9)
    Male: number analyzed (Participants) | 17
    Male | 37.3 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Subjective Overall Score
Description: Subjective overall score was assessed using 0-100 visual analogue scale, where 0=Extremely poor, cannot use lenses and 100=Excellent, highly impressed with these lenses overall
Time Frame: 15 minutes
Population: One participant was excluded from data analysis due to issues during lens application
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Lens 1: All participants that received Lens 1
- Lens 2: All participants that received Lens 2
Arm/Group | Lens 1 | Lens 2
Number analyzed (Participants) | 44 | 44
score on a scale | 84.7 (15.5) | 82.5 (14.6)

2. Secondary Outcome: Subjective Comfort
Description: Subjective comfort score was assessed using 0-100 visual analogue scale, where 0=Causes pain, cannot be tolerated and 100=Excellent, cannot be felt
Time Frame: 15 minutes
Population: One participant was excluded from data analysis due to issues during lens application
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lens 1 | Lens 2
Number analyzed (Participants) | 44 | 44
score on a scale | 86.4 (16.4) | 86.6 (13.5)

3. Secondary Outcome: Subjective Vision
Description: Subjective vision score was assessed using a 0-100 visual analogue scale, where 0=Unacceptable, lens cannot be worn and 100=Excellent, unaware of any visual loss
Time Frame: 15 minutes
Population: One participant was excluded from data analysis due to issues during lens application
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lens 1 | Lens 2
Number analyzed (Participants) | 44 | 44
score on a scale | 85.8 (14.9) | 82.7 (15.9)

ADVERSE EVENTS:
Time Frame: The duration of the clinical trial, approximately 1.5 hours
Arm/Group | Lens 1 | Lens 2
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/50/NCT05741450/Prot_SAP_000.pdf